CLINICAL TRIAL: NCT04484220
Title: Ellipsys Vascular Access System Post Market Surveillance (PS) Study PS200001 Reference DEN170004
Brief Title: Ellipsys Vascular Access System Post Market Surveillance (PS) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PS200001
Record Dates: First submitted 2020-06-25; First posted 2020-07-23 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Renal Disease, End Stage; Kidney Disease, End-Stage; AV Fistula; Fistulas Arteriovenous
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Ellipsys Vascular Access System (Experimental): The Ellipsys System is indicated for the creation of a proximal radial artery to perforating vein anastomosis via a retrograde venous access approach in patients who have chronic kidney disease requiring dialysis.
  Interventions: Device: Ellipsys Vascular Access System

INTERVENTIONS:
Device: Ellipsys Vascular Access System — The Ellipsys System is indicated for the creation of a proximal radial artery to perforating vein anastomosis via a retrograde venous access approach in patients with a minimum vessel diameter of 2.0mm and less than 1.5mm of separation between the artery and vein at the fistula creation site who have chronic kidney disease requiring dialysis.

SUMMARY:
The proposed clinical study is a prospective, non-randomized, multi-center, single-arm, observational, post-market surveillance (PS) study of the Ellipsys Vascular Access System in subjects eligible for arteriovenous (AV) fistula.

DETAILED DESCRIPTION:
The primary objective of this post-market surveillance study is to support the short-term safety of the device and procedure and further assess long-term safety and effectiveness in subjects treated by newly trained providers of the Ellipsys Vascular Access System in the creation of a native AV fistula via percutaneous access in subjects who are on hemodialysis and are medically indicated for the creation of an upper limb anastomosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female ≥ 18 years of age and ≤ 80 years of age
2. Life expectancy of at least one year, in the investigator's opinion
3. Diagnosed with ESRD or chronic kidney disease on hemodialysis.
4. Patients deemed medically eligible for upper extremity autogenous AV fistula creation, per institutional guidelines and/or clinical judgment
5. Adequate quality vein based on pre-operative assessment

   1. Adjacent vein diameter of ≥2.0 mm at target anastomosis site
   2. Confirmed clinically significant outflow
6. Adequate quality radial artery based on pre-operative assessment

   a. Arterial lumen diameter of ≥2.0 mm at target anastomosis site
7. Adequate collateral arterial perfusion with patent palmar arch as demonstrated by Barbeau Test or Allen's Test.
8. Radial artery-adjacent vein proximity ≤1.5 mm measured lumen edge-to-lumen edge as determined by pre-procedural ultrasound and confirmed pre-procedure
9. Patient is able to provide written informed consent and attend follow-up examinations at the enrolling institution

   Imaging-based Inclusion Criteria:
10. Confirm radial artery-adjacent vein proximity ≤1.5 mm measured lumen edge-to-lumen edge as determined by pre-procedural ultrasound and confirmed pre-procedurally
11. Confirm radial artery and adjacent vein diameter of ≥2.0 mm at target anastomosis site

Exclusion Criteria:

1. Pre-existing ipsilateral vascular disease interfering with the study procedure or potentially confounding the study results including:

   1. Documented or suspected central venous stenosis (≥ 50%) or
   2. Upper extremity arterial stenosis or
   3. Vascular disease at the radial artery / adjacent vein site
2. Prior vascular surgery at or proximal (central) to the AVF target site interfering with AVF maturation or other ipsilateral surgery that could potentially confound the study results such as prior axillary dissection or mastectomy
3. History of steal syndrome from a previous surgical ipsilateral hemodialysis vascular access which required intervention or abandonment
4. Systolic pressures < 100 mg Hg at the time of screening
5. Suspected or confirmed skin disease at the skin entry site
6. Edema of the upper extremity on the ipsilateral side
7. Immunocompromised subjects due to underlying disease or immunosuppressant therapy such as sirolimus (Rapamune®) or Prednisone at a dose of > 10 mg per day
8. Known bleeding diathesis, coagulation disorder or medications putting the subject at increased risk, in the Investigator's judgment
9. Patients with acute or active infection
10. Scheduled kidney transplant within 6 months of enrollment
11. Participation in another clinical investigation (excluding retrospective studies or studies not requiring a consent form)
12. History of substance abuse or anticipated to be non-compliant with medical care or study requirements based on investigator judgment
13. Patient has an active COVID-19 infection with ongoing sequela or hospitalization for treatment of COVID-19.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Cumulative Patency Through 12 months Post-AVF Creation | 12 months post-procedure
  Freedom from access abandonment from time of access creation
Early Occlusion Rate at 7 days | 7 days post-procedure
  Percent of patients with total occlusion within 7 days of the AVF creation procedure
Study Related Serious Adverse Event (SAE) Rate Through 12 months | 12 months post-procedure
  Rate of serious adverse events through 12 months related to the device, study procedure, or secondary procedure to maintain or re-establish patency.

SECONDARY OUTCOMES:
Primary Patency Through 12 months Post-AVF Creation | 12 months post-procedure
  Freedom from access thrombosis or any intervention designed to facilitate, maintain or re-establish patency measured from time of access creation through 12 months
Assisted Primary Patency Through 12 months Post-AVF Creation | 12 months post-procedure
  Freedom from access thrombosis from time of access creation
Secondary Procedures Rate | 12 months post-procedure
  Number of surgical or percutaneous interventions designed to mature or maintain the AVF or re-establish flow per person-year.
Overall Patient Safety | 12 months post-procedure
  A full characterization of adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Haimanot Wasse, MD, Principal Investigator — Rush University Medical Center
Locations (12):
- United States (12):
  - Nephrology Associates Access Center, Riverside, California
  - Yale University, New Haven, Connecticut
  - Azura Vascular Care, Jacksonville, Jacksonville, Florida
  - Coastal Vascular and Interventional, PLLC, Pensacola, Florida
  - Rush University Medical Center, Chicago, Illinois
  - The Vascular Care Group, Hyannis, Massachusetts
  - Nephrology Kidney Disease Hypertension Center, Las Vegas, Nevada
  - Staten Island Hospital, Staten Island, New York
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - STAR Vascular Access Center, San Antonio, Texas
  - San Antonio Kidney Disease Center, San Antonio, Texas
  - Richmond Vascular Center, North Chesterfield, Virginia

IPD SHARING:
Plan to Share IPD: No